CLINICAL TRIAL: NCT04992000
Title: Self-Care of Hypertension of Older Adults During COVID-19 Lockdown Period: A Randomized Controlled Trial
Brief Title: Self-Care of Hypertension Among Older Adults During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Khitam Alsaqer, Principle Investigator, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YDU/2020/76-997
Record Dates: First submitted 2021-07-29; First posted 2021-08-05 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
Keywords: self-care; hypertension; COVID-19; m-Health; Older adults
MeSH Terms: conditions — Hypertension; COVID-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-free app + PHN intervention (Experimental): The intervention group was received initial education, 4-free apps, and followed by PHN interventions.
  Education, app, and PHN intervention
  Interventions: Other: 4-free app + PHN intervention
- 4-free app alone (Experimental): The apps alone group received the initial education and the 4-free Apps.
  Interventions: Other: 4-free app + PHN intervention
- education (No Intervention): Standard care group received just the initial education.

INTERVENTIONS:
Other: 4-free app + PHN intervention — same mentioned in groups
  Arms: 4-free app + PHN intervention; 4-free app alone

SUMMARY:
This study aimed to examine the effects of a public health nursing intervention plus m-Health applications for hypertension management on enhancing the Self-care, systolic and diastolic blood pressure, and quality of life in older adults during the lockdown period in Jordan.

Study Hypothesis:

There are no differences between the three groups in:

H01 HTN self-care (SC-HI) score. H02 Health-related quality of life (SF-36) score. H03 The management of systolic and diastolic BP levels.

DETAILED DESCRIPTION:
COVID-19 pandemic has affected all health aspects and aggravated chronic diseases health disparities because it is more common among vulnerable populations such as seniors 1. Hypertension (HTN) is a long-term chronic disease, affects more than 1 billion people around the world 2. In Jordan, one-third of Jordanian adults are hypertensive 3, one study expected that the prevalence of hypertension in 2013 may increase 7.2% by 2030 4, the HTN deaths rate touched 5% of total deaths, ranks Jordan number 7 in the world, and ranks the HTN at number 6 of leading causes of death, after coronary heart disease and stroke, the first and second leading causes of death in Jordan 5. If high blood pressure is uncontrolled, HTN is the main contributor to heart failure, cardiovascular disease, stroke, kidney disease, and death 2.

Concurrent with COVID-19, care is compromised in the context of lockdown and social distancing. Patients with chronic illness at his time have the risk that they are not obtaining the necessary hospital care, and alternative solutions are required, such as improving patient's self-care of his or her chronic disease 6. Since the hospitals are occupied with COVID-19 cases, the elderly have a perceived threat of COVID-19 and have begun avoiding or delaying health care follow-up 1. It is essential that the investigators find innovative solutions and sustainable methods for patients with HTN to control the blood pressure (BP), enhance self-care, and protect them from COVID-19, and ultimately improve their quality of life.

Engaging the patient in self-care makes him/her an active participant in the management of illness 7. Researchers worked to provide patients with the essential knowledge, skills and abilities to follow treatment recommendations and tolerate blood pressure control 8,9. Although they agreed that the best ways to prevent and manage high BP are through reasonable lifestyle changes, i.e., weight loss, low salt diet, stop smoking, limited alcohol, stress management, exercise, and medication 8, this makes the managing of high BP neither more difficult, nor easier.

However, to support healthy behaviors, the big electronic revolution provides a good opportunity to involve patients suffering from HTN in the health care process and self-care engagement in a safe space 10,11. Moreover, in order to adapt to disruptions during COVID-19, telehealth, mobile health (m-health), and other technologies which support the self-care process and facilitate access to care are appropriate approaches to protect vulnerable populations who are living with chronic diseases 1,12,13. However, improving the self-care of HTN using m-health is not a new approach; it has been studied previously by researchers from different disciplines such as technical medicine, family medicine, and pharmacy 14-19, with less attention given to the nursing role.

In literature, especially nursing literature, there is a lack of sufficient scientific research on the effectiveness of m-Health, guided by nurse's intervention, on self-care of HTN, particularly among older adults12,13. Recently, one study provided a nurse-led program as an example of an effective method to HTN management among older adults 20. The consequences of the COVID-19 pandemic (isolation, social distancing, quarantine) show major challenges in provision of care for older adults with chronic illness 1,6. The m-Health offers a great chance for providing care during the lockdown period, which can be applied via mobile apps 21. Thus, examining m-Health Apps guided by public health nursing (PHN) interventions for the management of HTN in older adults during the pandemic can provide important empirical evidence of effectiveness of such new innovative self-care of HTN interventional methods.

In this study, the investigators aim to examine three patients outcomes; self-care of HTN, change of systolic and diastolic of BP, and quality of life in three groups of older adult patients with HTN: the interventional group (4-free Apps + PHN interventions + education), control groups 1 (4-free Apps + education), and control group 2 (education) during the imposition of lockdown in Jordan as a result of COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were 55 years and above,
2. have follow-up with out-patients of KAUH,
3. had been diagnosed with hypertension,
4. on anti-hypertension medication- at least one drug,
5. reported that he/she has a personal smartphone (Android) - internet access is not important,
6. able to read and understand the Arabic language.

Exclusion Criteria:

1. Participants have Apple phones,
2. had any psychiatric or mental illness,
3. had a terminal-stage disease or were blind or deaf.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Self-care (SC-HI) scale | basic and after 3 months
  Self-care of HTN was measured by the SC-HI scale, which developed to measure the self-care in patients with HTN 26. SC-HI has the ability of evaluate the effectiveness of such self-care interventions. SC-HI is 23-item in three subscales: measuring self-care maintenance, monitoring, and management, Cronbach's α were 0.83, 0.75, and 0.83 for the three subscales. For the purpose of this study, authors cross-culturally translated the scale into Arabic in a previous study; Cronbach's α were 0.82, 0.61, and 0.86 for the three subscales 27. . Each subscale is scored distinctly and identical from 0 to 100, the final score calculated as: (the participant score - minimum) / (maximum - minimum) * 100. The separate score 70 or greater is indicated better self-care.
Changing in systolic and diastolic blood pressure | basic and after 3 months
  Systolic BP (SBP) and diastolic BP (DBP) were measured and recorded by a clinic nurse who has 9 years' experience in the cardiac clinic two times for the purpose of study's analysis; at baseline and after 3 months following the same assessment process: Patients in setting position with their arms at the chest line, relaxed for 5 minutes, then measuring the BP of the right arm using an electronic sphygmomanometer which was checked for calibrated regularly. BP readings through the 3 months were measured by patients themselves at home.

SECONDARY OUTCOMES:
Quality of life (SF-36) scale | basic and after 3 months
  Quality of life (QOL) of hypertensive patients was measured using the 36-Item Short Form Survey (SF-36). SF-36 questionnaire has been used as health indicator to screen the health status of persons and evaluate the health interventions 28. The questionnaire has the feasibility to be administered as a self-report, personal interview or by telephone, and takes 5-10 minutes to complete. SD-36 included 8 subscales: physical functioning (PF), bodily pain, role limitations due to physical health problems (RF), role limitations due to personal or emotional problems (RE), emotional well-being (EW), social functioning (SF), energy/fatigue (EF), and general health perceptions 28. SF-36 was frequently used to measure QOL in older adults with hypertension; the Arabic version was used in studies with Cronbach's α ≥ 0.70 29,30.

CONTACTS AND LOCATIONS:
Overall Officials: hatice Bebis, Prof. Dr, Principal Investigator — Near East University
Locations (1):
- Near east University, Nicosia, Cyprus

REFERENCES:
- [Derived] Alsaqer K, Bebis H. Self-care of hypertension of older adults during COVID-19 lockdown period: a randomized controlled trial. Clin Hypertens. 2022 Jul 15;28(1):21. doi: 10.1186/s40885-022-00204-7. PMID 35836287